CLINICAL TRIAL: NCT02465502
Title: An Uncontrolled, Open-label Phase IIb Trial of Regorafenib in Subjects With Antiangiogenic-naive and Chemotherapy-refractory Advanced Colorectal Cancer
Brief Title: Regorafenib in Subjects With Antiangiogenic-naive and Chemotherapy-refractory Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17217
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer; Regorafenib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib (BAY73-4506) (Experimental): Regorafenib 160 mg orally once a day for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off).
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib 160 mg orally once a day for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off).

SUMMARY:
To determine the efficacy (as measured by progression-free survival [PFS] rate at 8 weeks) of regorafenib in subjects with metastatic colorectal cancer (CRC) whose disease is refractory to standard therapies and who were never exposed to antiangiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age;
* Histological or cytological confirmation of adenocarcinoma of the colon or/and rectum;
* Subjects with metastatic colorectal cancer (CRC) whose disease progressed or who were intolerant to standard chemotherapy based on fluoropyrimidine, oxaliplatin, irinotecan, and an anti-EGFR therapy if RAS wild-type. This progression must be during or within 4 months following the last administration of standard therapies.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone-marrow, liver, and renal function
* Women of childbearing potential and men must agree to use adequate contraception when sexually active during the study and for at least 8 weeks after the last study drug administration.

Exclusion Criteria:

* Prior treatment with an antiangiogenic agent;
* Congestive heart failure of New York Heart Association (NYHA) class 2 or worse;
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study drug;
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg despite optimal medical management);
* Ongoing acute or chronic infection (> Grade 2 NCI-CTCAE v 4.03);
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication) events within 6 months of study enrollment. Subjects being treated with low-weight heparin are allowed to participate as long as dose is limited to prophylactic use.
* Any history of or currently known brain metastases (head CT/MRI will be performed during screening period if brain metastases are suspected)
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years before study entry, except for curatively treated cervical cancer in situ, in situ ductal breast cancer, non-melanoma skin cancer and superficial bladder tumors;
* Last chemotherapy dose or any other anti-cancer therapy administered in less than 4 weeks from start of study treatment;
* Use of therapeutic anticoagulation;
* Proteinuria > 3.5 g/24 hours measured by urine protein-creatinine ratio from a random urine sample (Grade 3, NCI-CTCAE v 4.03) on urinalysis screening result. If there is medical history of proteinuria, previous urinalysis results should be considered and/or performed so at least 2 results separated by at least 2 weeks are available;
* History of interstitial lung disease with ongoing signs and symptoms at the time of informed consent;
* Non-healing wound, non-healing ulcer, or non-healing bone fracture;
* Subjects with evidence or history of any bleeding diathesis, irrespective of severity;
* Any hemorrhage or bleeding event ≥ Grade 3 NCI-CTCAE v 4.03 within 4 weeks prior to the start of study medication;
* Known history of human immunodeficiency virus (HIV) infection;
* History of active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy;
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants without disease progression or death at the end of 8 weeks | At week 8

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 2 months
  PFS is defined as the date from the first dose of regorafenib until radiologic and/or clear clinical progression or death from any cause, whichever comes first.
Overall Survival (OS) | Approximately 2 months
  OS is defined as the date from the first dose of regorafenib until death by any cause.
Overall Response Rate (ORR) | Approximately 2 months
  ORR is defined as the proportion of subjects with the best tumor response (confirmed PR or CR) that is achieved during or within 30 days after therapy.
Disease Control Rate (DCR) | Approximately 2 months
  DCR is defined as the proportion of subjects who have a best response rating over the whole duration of the study of CR, PR, or SD.
Metabolic response measured by [18F] fluorodeoxyglucose positron emission tomography (FDG PET) | Approximately 2 months
Percentage of participants with grade 1 or higher adverse events, using NCI Common Terminology Criteria for Adverse Events (CTC-AE) Version 4.03 | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- São Paulo, Brazil

REFERENCES:
- [Derived] Riechelmann RP, Leite LS, Bariani GM, Glasberg J, Rivelli TG, da Fonseca LG, Nebuloni DR, Braghiroli MI, Queiroz MA, Isejima AM, Kappeler C, Kikuchi L, Hoff PM. Regorafenib in Patients with Antiangiogenic-Naive and Chemotherapy-Refractory Advanced Colorectal Cancer: Results from a Phase IIb Trial. Oncologist. 2019 Sep;24(9):1180-1187. doi: 10.1634/theoncologist.2019-0067. Epub 2019 Jun 7. PMID 31175167